CLINICAL TRIAL: NCT00962832
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rontalizumab (rhuMAb IFNalpha) in Patients With Moderately to Severely Active Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Rontalizumab in Patients With Moderately to Severely Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFN4575g; GA00806 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: rhuMAb IFNalpha; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — rontalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Part 1 - Placebo intravenously (Placebo Comparator): Participants received placebo intravenously every 4 weeks for 24 weeks.
  Interventions: Drug: Placebo
- Part 1 - Rontalizumab 750 mg intravenously (Experimental): Participants received rontalizumab 750 mg intravenously every 4 weeks for 24 weeks.
  Interventions: Drug: Rontalizumab
- Part 2 - Placebo subcutaneously (Placebo Comparator): Participants received placebo subcutaneously every 2 weeks for 24 weeks.
  Interventions: Drug: Placebo
- Part 2 - Rontalizumab 300 mg subcutaneously (Experimental): Participants received rontalizumab 300 mg subcutaneously every 2 weeks for 24 weeks.
  Interventions: Drug: Rontalizumab
- Part 3 - Rontalizumab 750 mg intravenously (Experimental): Participants received rontalizumab 750 mg intravenously every 4 weeks for 120 weeks.
  Interventions: Drug: Rontalizumab

INTERVENTIONS:
Drug: Placebo — Placebo was supplied as a sterile liquid solution.
  Arms: Part 1 - Placebo intravenously; Part 2 - Placebo subcutaneously
Drug: Rontalizumab — Rontalizumab was supplied as a sterile liquid solution.
  Arms: Part 1 - Rontalizumab 750 mg intravenously; Part 2 - Rontalizumab 300 mg subcutaneously; Part 3 - Rontalizumab 750 mg intravenously

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of rontalizumab compared with placebo in patients with moderately to severely active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
The study will be conducted in 3 parts. Parts 1 and 2 of the study will include a double-blind treatment period of 24 weeks and a safety follow-up period of 48 weeks for participants who do not continue onto Part 3. Patients meeting the eligibility criteria for enrollment in Part 3, will enter Part 3 after completion of the Week 24 visit but prior to completion of the Week 72 visit. In Part 1, participants will be randomized in a 2:1 ratio (active drug:placebo) to receive either rontalizumab 750 mg or matching placebo intravenously every 4 weeks for 24 weeks. Part 2 was will be initiated upon the completion of recruitment for Part 1. In Part 2, participants will be randomized in a 2:1 ratio (active drug:placebo) to receive either rontalizumab 300 mg or matching placebo subcutaneously every 2 weeks for 24 weeks. After Week 24, patients will enter a 48-week safety follow-up period, or, after the open label extension became available via protocol amendment, will have the option of entering Part 3 of the study, if eligible. In Part 3, all participants will receive rontalizumab 750 mg intravenously every 4 weeks for 120 weeks (up to 144 weeks total).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE.
* Active disease at the time of screening.
* Agreement to use an effective form of contraception for the duration of the study.

Exclusion Criteria:

* Acutely life- or organ-threatening manifestations of systemic lupus erythematosus (SLE) (eg, proliferative nephritis, unstable neuropsychiatric disease).
* Pregnancy or breastfeeding.
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or intravenous (IV) immunoglobulin.
* Significant, uncontrolled medical disease in any organ system not related to SLE that in the investigator's opinion would preclude patient participation.
* Concomitant conditions that required systemic corticosteroid use within 1 year prior to screening. Use of topical, intraarticular, or inhaled corticosteroids is not exclusionary.
* History of cancer within 5 years of screening.
* Any current or recent (within 4 weeks of screening) signs or symptoms of infection, except for minor infections, fungal infections of the nail beds, or oral or vaginal candidiasis.
* History of severe systemic bacterial, fungal, viral, or parasitic infections (2 or more hospitalizations or 2 or more courses of IV antibiotics) within 6 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of responders at Week 24 | Until study discontinuation or up to 24 weeks

SECONDARY OUTCOMES:
Time-adjusted area under the curve (AUC) of the BILAG index global score | Until study discontinuation or up to 24 weeks
Treatment failure status | Until study discontinuation or up to 24 weeks
Time to treatment failure | Until study discontinuation or up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Kennedy, M.D., Study Director — Genentech, Inc.
Locations (72):
- United States (43):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Tucson, Arizona
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - San Leandro, California
  - Upland, California
  - Aventura, Florida
  - Clearwater, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Kansas City, Kansas
  - Baton Rouge, Louisiana
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Brooklyn, New York
  - Great Neck, New York
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Roslyn, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Sugar Land, Texas
  - Arlington, Virginia
  - Spokane, Washington
- Argentina (4):
  - Buenos Aires
  - Ciudad Autonoma Buenos A.
  - Rosario
  - San Miguel de Tucumán
- Colombia (7):
  - Barranquilla
  - Barranquilla-Atlantico
  - Bogota D.C.
  - Bogotá
  - Bucaramanga
  - Chia-Cundinamarca
  - Medellin-Antioquia
- Mexico (7):
  - Guadalajara
  - Mexico City
  - Mexico Ctiy
  - México
  - Miexico City
  - Morelia
  - San Luis Potosi S.l.p.
- Poland (7):
  - Bydgoszcz
  - Elblag
  - Gmina Końskie
  - Kościan
  - Krakow
  - Poznan
  - Warsaw
- Russia (4):
  - Kazan'
  - Moscow
  - Tomsk
  - Yaroslavl

REFERENCES:
- [Derived] Kalunian KC, Merrill JT, Maciuca R, McBride JM, Townsend MJ, Wei X, Davis JC Jr, Kennedy WP. A Phase II study of the efficacy and safety of rontalizumab (rhuMAb interferon-alpha) in patients with systemic lupus erythematosus (ROSE). Ann Rheum Dis. 2016 Jan;75(1):196-202. doi: 10.1136/annrheumdis-2014-206090. Epub 2015 Jun 2. PMID 26038091
- [Derived] Kennedy WP, Maciuca R, Wolslegel K, Tew W, Abbas AR, Chaivorapol C, Morimoto A, McBride JM, Brunetta P, Richardson BC, Davis JC Jr, Behrens TW, Townsend MJ. Association of the interferon signature metric with serological disease manifestations but not global activity scores in multiple cohorts of patients with SLE. Lupus Sci Med. 2015 Mar 28;2(1):e000080. doi: 10.1136/lupus-2014-000080. eCollection 2015. PMID 25861459